CLINICAL TRIAL: NCT01691105
Title: Implementation of HIT-Enhanced Tobacco Treatment for Hospitalized Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1205010297; R18HL108788 (NIH)
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Tobacco Use Cessation; Smoking Cessation; Smoking; Tobacco Use Disorder
Keywords: Tobacco Use Cessation; Smoking Cessation; Nicotine Replacement Therapy; Hospitalized Smokers
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation; Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Academic Detailing (AD) (No Intervention): Standard of care for patients who are smokers and admitted to the hospital.
- AD + Integrated Tobacco Order Set (Experimental): Access to the Integrated Tobacco Order Set (ITOS) Nicotine Replacement Therapy with dosing instructions Bupropion and varenicline with dosing instructions Automated referral to the CT Quitline Automated fax to PCP Discharge prescription prompt Quitline report sent to PCP 2 day call back from hospital call center
  Interventions: Other: AD + Integrated Tobacco Order Set

INTERVENTIONS:
Other: AD + Integrated Tobacco Order Set — Physician will have access to:
  NRT with dosing instructions Bupropion and varenicline with dosing instructions Automated referral to the CT Quitline Automated fax to PCP Discharge prescription prompt Quitline report sent to PCP 2 day call back from hospital call center
  Arms: AD + Integrated Tobacco Order Set

SUMMARY:
This study will implement and test the effectiveness and cost-effectiveness of a tobacco cessation intervention (Academic Detailing + Integrated Tobacco Order Set - AD + ITOS) for adults admitted to the hospital. The intervention will begin during the hospital stay and continue after discharge. The intervention will use resources easily available to most acute care hospitals: computerized physician order entry, physician and nurse education, staff meetings for physicians, nurses and allied health professionals, online learning capabilities, faxing to primary care providers (PCPs), and the telephone counseling and support available from a state smokers' quitline (QL).

The investigators hypothesize that the subjects in the intervention arm (AD + ITOS) will be more likely to achieve tobacco abstinence at 12 months post hospital stay than subjects in the control arm (Academic Detailing - AD). Tobacco abstinence will be assessed by self report and biochemical verification (exhaled carbon monoxide reading).

DETAILED DESCRIPTION:
Cigarette smoking remains the leading cause of preventable death and illness in the United States. In 2008, 20.6% of all American adults smoked, and 435,000 died from smoking-related illnesses. Economic costs of smoking dependence are estimated at $193 billion/year and have far-reaching implications for the individual, workplace, society and the healthcare system. However, treatment is associated with significant individual and society benefits, and both counseling and pharmacotherapy have been demonstrated to be effective treatments. Along with poverty and low education, smoking causes a greater loss of quality-adjusted life years than race, uninsurance, overweight, or binge drinking.

Smokers are admitted to acute care hospital more than nonsmokers. Using estimates from a number of sources, we estimate that approximately 6.1-12.5 million hospitalizations occur annually among adult smokers. This represents 20-41% of the 29.8 million annual inpatient stays in US acute care hospitals among adults age 18 and older unrelated to pregnancy or childbirth. Put another way, the nation's 46 million smokers represent 20% of the adult population, but account for 20-40% of all hospitalizations unrelated to pregnancy. Given that US hospitals are now smoke-free (per Joint Commission regulations), and many of these admissions are for tobacco-related conditions, the hospital admission represents a profound opportunity-a "teachable moment"-for tobacco control.

Recent "core measure" regulations by the Joint Commission and the Centers for Medicare and Medicaid Services require hospitals to report publicly their tobacco screening for patients admitted with acute myocardial infarction, congestive heart failure, and pneumonia. Although many hospitals have improved their performance considerably on these smoking measures, sometimes this has resulted from "gaming," e.g. giving all discharged patients a preprinted instruction sheet that includes boilerplate text about smoking cessation. Thus, although most hospitals assess inpatients for tobacco use (either through a nursing assessment or the physician's initial history and physical examination), there are often no systems in place to initiate or sustain tobacco treatment for smokers. This gap in service delivery prevents millions of smokers from accessing the many effective, evidence-based treatments for tobacco dependence during a period in which they may be particularly receptive to an intervention.

Hence, the overarching goal of this project is to implement and study the effectiveness and cost-effectiveness of a tobacco intervention for hospitalized adults that begins during inpatient treatment and continues after discharge. To enhance dissemination, we will use resources currently available to most acute care hospitals: computerized physician order entry, physician and nurse education, staff meetings for physicians, nurses, and allied health professionals, online learning capabilities, faxing to primary care providers (PCPs), and the telephone counseling and support available from a state smokers' quitline (QL). In the final year, a toolkit will be disseminated by professional societies. We hypothesize that the proposed intervention is clinically effective, cost effective, sustainable, and generalizable. All interventions are evidence-based and consistent with the 2008 Public Health Service clinical practice guideline for tobacco dependence treatment.

The Specific Aims of the proposed project are to:

Primary Aims:

1. Determine whether Academic Detailing (AD) and an Integrated Tobacco Order Set (ITOS) compared to AD alone improves biologically verified smoking cessation at 12 months post-quit in a cohort of 960 smokers age > 18 years admitted to Yale New Haven Hospital (YNHH).

   Secondary Aims:
2. Study ITOS's ability to encourage smokers to use treatment services and reduce consumption.
3. Study ITOS's ability to enhance provider delivery of tobacco screening and treatment.
4. Conduct an incremental cost-effectiveness analysis of the intervention.

Our associated hypotheses are:

1. Subjects treated by physicians in the AD+ITOS arm will have a higher rate of biochemically verified 7-day point prevalence smoking abstinence at 12 months post-quit than subjects treated by physicians in the AD arm, in a cohort of adult smokers admitted to the inpatient units of Yale-New Haven Hospital.
2. Subjects treated by AD+ITOS physicians will have made more quit attempts, and experienced greater reduction in daily cigarette consumption, than smokers treated by AD physicians.
3. A higher proportion of patients treated by AD+ITOS physicians will have tobacco treatment initiated in hospital than patients treated by AD physicians.
4. Societal costs of AD+ITOS, per abstinent smoker, will be cost-effective relative to AD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* admitted to any medical ward, telemetry or cardiac care unit
* identified as a smoker by the nurse or physician in the admitting EMR
* treated by a study physician
* able to give written informed consent

Exclusion Criteria:

* inability to read or understand English or Spanish
* lacks capacity to give informed consent
* currently receiving formal tobacco dependence treatment
* current suicide or homicide risk
* current psychotic disorder or life-threatening or unstable medical or psychiatric condition within past 6 months
* unable to provide 2 telephone contact numbers
* unwilling to follow up per study protocol, including release of information to assess treatment engagement at 30-days
* live outside of New Haven County
* leaving the hospital against medical advice
* history of clinically significant allergic reaction to nicotine replacement therapies, varenicline or bupropion
* use of an investigational drug within 30 days
* use of tobacco products other than cigarettes
* women of childbearing potential who are pregnant, nursing, or sexually active and not practicing effective contraception (oral injectable, or implantable contraceptives, intrauterine device, or barrier method with spermicide)
* do not have access to a phone with a CT area code (required to use the CT Tobacco Quitline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Bernstein, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Bernstein SL, Weiss J, DeWitt M, Tetrault JM, Hsiao AL, Dziura J, Sussman S, Miller T, Carpenter K, O'Connor P, Toll B. A randomized trial of decision support for tobacco dependence treatment in an inpatient electronic medical record: clinical results. Implement Sci. 2019 Jan 22;14(1):8. doi: 10.1186/s13012-019-0856-8. PMID 30670043
- [Derived] Bernstein SL, Rosner J, DeWitt M, Tetrault J, Hsiao AL, Dziura J, Sussman S, O'Connor P, Toll B. Design and implementation of decision support for tobacco dependence treatment in an inpatient electronic medical record: a randomized trial. Transl Behav Med. 2017 Jun;7(2):185-195. doi: 10.1007/s13142-017-0470-8. PMID 28194729

RESULTS

PARTICIPANT FLOW:
Groups:
- AD + Integrated Tobacco Order Set: Access to the Integrated Tobacco Order Set (ITOS) Nicotine Replacement Therapy with dosing instructions Bupropion and varenicline with dosing instructions Automated referral to the CT Quitline Automated fax to PCP Discharge prescription prompt Quitline report sent to PCP 2 day call back from hospital call center
  AD + Integrated Tobacco Order Set: Physician will have access to:
  NRT with dosing instructions Bupropion and varenicline with dosing instructions Automated referral to the CT Quitline Automated fax to PCP Discharge prescription prompt Quitline report sent to PCP 2 day call back from hospital call center
Period: Baseline
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Started | 477 | 567
Completed | 477 | 567
Not Completed | 0 | 0
Period: 1 Month Follow-up
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Started | 477 | 567
Completed | 434 | 526
Not Completed | 43 | 41
Not completed — Lost to Follow-up | 41 | 38
Not completed — Death | 2 | 3
Period: 6 Month Follow-up
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Started | 477 | 567
Completed | 425 | 496
Not Completed | 52 | 71
Not completed — Lost to Follow-up | 39 | 58
Not completed — Death | 13 | 13
Period: 12 Month Follow-up
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Started | 477 | 567
Completed | 405 | 466
Not Completed | 72 | 101
Not completed — Lost to Follow-up | 50 | 71
Not completed — Death | 22 | 30
Period: 12 Month Biochemical Verification
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Started | 477 | 567
Completed | 53 | 65
Not Completed | 424 | 502
Not completed — Death | 22 | 30
Not completed — Lost to Follow-up | 50 | 71
Not completed — subject did not self-report abstinence | 352 | 401

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set | Total
Number analyzed (Participants) | 477 | 567 | 1044
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (12.6) | 49.3 (11.7) | 49.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 286 | 524
  Male | 239 | 281 | 520
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 61 | 112
  Not Hispanic or Latino | 426 | 506 | 932
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 157 | 170 | 327
  White | 303 | 372 | 675
  More than one race | 11 | 18 | 29
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 477 | 567 | 1044
Cigarettes/day [Median (Inter-Quartile Range); unit: cigarettes per day] | 10.0 [8 to 20] | 10.5 [8 to 20] | 10.0 [8 to 20]
Heavy Smoking Index >= 4, N (%) [Count of Participants; unit: Participants] | 208 | 210 | 418

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Exhaled Carbon Monoxide Confirmed Abstinence
Description: Tobacco abstinence will be assessed by obtaining an exhaled carbon monoxide reading for all subjects self-reporting tobacco abstinence at 12 month follow-up. Consistent with manufacturer's recommendations, a cutoff of 10 ppm will indicate current smoking.
Time Frame: 12 months post enrollment
Population: Only participants self-reporting abstinence during the 12 month follow-up call were asked to provide biochemical verification.
Measure: Number; unit: participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 78 | 86
participants | 53 | 65

2. Secondary Outcome: Number of Participants With Self-Reported Tobacco Reduction or Abstinence - 12 Months
Description: Self-report questionnaires are completed over the phone to assess reduction in cigarette use or abstinence from cigarette use. The Time Line Follow Back technique will be used to assess 7-day point prevalence abstinence.
Time Frame: 12 months post enrollment
Population: Only includes participants who completed the 12 month follow-up appointment.
Measure: Number; unit: participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 405 | 466
participants | 78 | 86

3. Secondary Outcome: Number of Participants With Self-Reported Tobacco Reduction or Abstinence - 6 Months
Description: as for outcome 2
Time Frame: 6 months post enrollment
Population: Includes only participants who completed the 6 month follow-up appointment.
Measure: Number; unit: participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 425 | 496
participants | 68 | 83

4. Secondary Outcome: Number of Participants With Self-Reported Tobacco Reduction or Abstinence - 1 Month
Description: as for outcome 2
Time Frame: 1 month post enrollment
Population: Includes only participants who completed 1 month follow-up appointment.
Measure: Number; unit: participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 434 | 526
participants | 72 | 87

5. Secondary Outcome: Number of Participants Self-Reporting Use of Cessation Medications - 1 Month
Description: Nicotine replacement therapy (NRT) use and use of other pharmacotherapies will be assessed by self-report. A Treatment Services Review (TSR) will be administered during follow-up assessments at 1, 6, and 12 months post enrollment.
Time Frame: 1 month post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 434 | 526
Participants | 126 | 187

6. Secondary Outcome: Number of Participants Self-Reporting Use of Cessation Medications - 6 Months
Description: NRT use and use of other pharmacotherapies will be assessed by self-report. A Treatment Services Review (TSR) will be administered during follow-up assessments at 6 months post enrollment.
Time Frame: 6 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 425 | 496
Participants | 100 | 146

7. Secondary Outcome: Number of Participants Self-Reporting Use of Cessation Medications - 12 Months
Description: NRT use and use of other pharmacotherapies will be assessed by self-report. A Treatment Services Review (TSR) will be administered during follow-up assessments at 1, 6, and 12 months post enrollment.
Time Frame: 12 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 405 | 466
Participants | 100 | 136

8. Secondary Outcome: Number of Participants Self-Reporting Treatment Engagement - 1 Month
Description: Treatment engagement will be assessed by subject self-report during the 1 month follow-up interview. Subjects will be considered engaged in treatment if at 30 days after randomization the subject reports currently receiving care for the Quitline or another treatment program that addresses the subject's nicotine dependence.
Time Frame: 1 month post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
Number analyzed (Participants) | 434 | 526
Participants | 32 | 80

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Academic Detailing (AD) | AD + Integrated Tobacco Order Set
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No